CLINICAL TRIAL: NCT04354194
Title: Osteopathic Manipulative Treatment in Chronic Non-specific Neck Pain: A Controlled Study
Brief Title: Osteopathic Manipulative Treatment in Chronic Non-specific Neck Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Şule (Other)
Responsible Party: Sponsor-Investigator, Şule, Principal Investigator, Pamukkale University
Organization: Pamukkale University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21.05.2019/10
Record Dates: First submitted 2020-04-13; First posted 2020-04-21 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Chronic Pain
Keywords: Osteopathic Manipulative Treatment; Chronic Non-spesific Neck Pain; Conventional Therapy
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Physiotherapy Group (Experimental): This group will receive 15 sessions of conventional physiotherapy programme 5 times per week.
  Interventions: Procedure: Conventional Physiotherapy
- Osteopathic Manipulative Treatment Group (Experimental): This group will receive 9 sessions of Osteopathic Manipulative Treatment programme 3 times per week.
  Interventions: Procedure: Osteopathic Manupilative Treatment

INTERVENTIONS:
Procedure: Conventional Physiotherapy — Conventional Physiotherapy consist of Hotpacks, TENS and US.The participants were positioned in sitting and supported with a pillow under the head, 20 min hot pack was applied. Therapatic Ultrason were applied with the frequency of 1 MHz, intensity of 1,5 watt/cm² and duration of 5 minute. TENS was applied to the cervical region with 2-channel, 4 surface electrodes at 60-120 Hz, and 50-100 pulse duration for 20 minutes.
  Arms: Conventional Physiotherapy Group
Procedure: Osteopathic Manupilative Treatment — Osteopathic Manupilative Treatment consist of stretching the fascia to the cervical region, soft tissue mobilization to the surrounding muscles, cervical manual traction, passive joint mobilization to the 7 cervical spine, passive joint mobilization to the 1st costa, passive joint mobilization to the clavicle and passive joint mobilization to the sternum mobilization in supine and prome positions.
  Arms: Osteopathic Manipulative Treatment Group

SUMMARY:
The aim of this study is to investigate the effect of osteopathic manipulative treatment on pain intensity, disability level and psychosocial factors in patients with chronic non-specific neck pain. We hypothesed that osteopathic manipulative treatment is better than conventional physiotherapy in management of pain, disability and depression.

DETAILED DESCRIPTION:
This study will conduct between April 2020 and July 2020 at Denizli State Hospital. Participants who were diagnosed as chronic non-specific neck pain by a specialist physician will include the study. They will treated at physical therapy clinic. Inclussion criteria will; participants diagnosed as non-specific neck pain by the physician and Non-spesific neck pain at least 3 months. Exclussion criteria were; participants who have had surgery or are indicated for surgery, participants who have had exercise therapy and / or physical therapy in the last 1 year with a history of trauma to the cervical region, participants who have had neck pain that develop due to a particular cause such as tumor, compression fracture, metastasis and infection. According to power analysis, 102 participant will include the study with 95% coincidence interval and 80% power. Participants will be divided into 2 groups. Randomization method will be closed envelope. Group 1 will receive Conventional Physiotherapy Programme (CP), Group 2 will receive Osteopathin Manipulative Treatment (OMT). Pain Intensity at rest and activity, psychological state( Beck Depression Inventory) and Disability level (Neck Disability Index) will assess at baseline and 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

* participants diagnosed as non-specific neck pain by the physician.
* Non-spesific neck pain at least 3 months.

Exclusion Criteria:

* participants who have had surgery or are indicated for surgery
* participants who have had exercise therapy and / or physical therapy in the last 1 year with a history of trauma to the cervical region
* participants who have had neck pains that develop due to a particular cause such as tumor, compression fracture, metastasis and infection

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2020-09-20 (Estimated); Study Completion 2020-12-20 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity | Change from baseline pain intensity at 3 weeks
  pain intensity at rest and activity will measure by VAS

SECONDARY OUTCOMES:
Disability level | Change from baseline Neck Disability Index score at 3 weeks
  Disability level will measue by Neck Disability Index. Score ranges from 0-100. Higher score indicates worse outcome.
Depression level | Change from baseline Beck Depression Inventory score at 3 weeks
  Depression will measure by Beck Depression Inventory. Scores ranges from 0-63. Higher score indicates worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Nesrin Yağcı, Prof., Study Director — Pamukkale University
Locations (1):
- Denizli State Hospital, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Because there is no web site to share my data

REFERENCES:
- [Background] Schwerla F, Bischoff A, Nurnberger A, Genter P, Guillaume JP, Resch KL. Osteopathic treatment of patients with chronic non-specific neck pain: a randomised controlled trial of efficacy. Forsch Komplementmed. 2008 Jun;15(3):138-45. doi: 10.1159/000132397. Epub 2008 Jun 4. PMID 18617745
- [Background] Jarski RW, Loniewski EG, Williams J, Bahu A, Shafinia S, Gibbs K, Muller M. The effectiveness of osteopathic manipulative treatment as complementary therapy following surgery: a prospective, match-controlled outcome study. Altern Ther Health Med. 2000 Sep;6(5):77-81. PMID 10979164
- [Background] Edwards DJ, Toutt C. An evaluation of osteopathic treatment on psychological outcomes with patients suffering from chronic pain: A prospective observational cohort study collected through a health and well-being academy. Health Psychol Open. 2018 May 10;5(1):2055102918774684. doi: 10.1177/2055102918774684. eCollection 2018 Jan-Jun. PMID 29780605
- [Result] Verhaeghe N, Schepers J, van Dun P, Annemans L. Osteopathic care for low back pain and neck pain: A cost-utility analysis. Complement Ther Med. 2018 Oct;40:207-213. doi: 10.1016/j.ctim.2018.06.001. Epub 2018 Jun 9. PMID 30219451